CLINICAL TRIAL: NCT01349530
Title: Evaluating of the Benefit to the Patient by Managing of His Anticoagulation Treatment by an Anti-coagulation Clinic
Brief Title: Evaluating of CREATIF an Anti-coagulation Clinic
Acronym: CREATIF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Ministry of Health, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: K080905; 2010-A00213-36 (Other: IDRCB)
Record Dates: First submitted 2011-05-05; First posted 2011-05-06 (Estimated); Last update posted 2017-01-04 (Estimated); Status verified 2016-12

CONDITIONS: Vitamin K Antagonist
Keywords: Usual medical care; Anticoagulation by VKAs: COUMADINE® & PREVISCAN®; Anticoagulation clinic care, CREATIF

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Anticoagulation clinic care (Experimental): Monitoring by CREATIF
  Interventions: Other: Evaluation of CREATIF
- Usual care (Active Comparator): Monitoring by GP.
  Interventions: Other: Evaluating of usual care

INTERVENTIONS:
Other: Evaluating of usual care — RESEARCH IN CURRENT CARE
  Arms: Usual care
Other: Evaluation of CREATIF — RESEARCH IN CURRENT CARE
  Arms: Anticoagulation clinic care

SUMMARY:
Main objective: To evaluate the impact of CREATIF (an anticoagulation clinic in Ile de France) on monitoring and management of patients treated with VKAs compared with usual primary care.

Study hypothesis: The investigators suppose that patients will have a better quality of anticoagulation when they are managed by CREATIF than by their usual General Physicians (GP)

DETAILED DESCRIPTION:
Vitamin K antagonists (VKA) are the reference of anticoagulant oral therapy concerning common diseases such as Atrial Fibrillation (AF) and Venous ThromboEmbolism (VTE). In France, approximately 600,000 patients are treated with oral anticoagulants. The treatment is monitored and adjusted on the INR. Time outside the area of target INR is directly correlated with complications (thrombotic and hemorrhagic), the time in this zone mean the effectiveness of treatment. In France, monitoring patients by GP, the percentage of the time outside the target area INR higher than their European or North American comparators. To reduce complications VKA, specialized structures for monitoring anticoagulation have emerged in recent years around the world (Netherlands, Italy, UK, Canada, and USA). The evaluations in these countries show that the percentage of time in therapeutic INR range is around 70% when the patient is monitored in anticoagulation clinic (ACC), while in France this time was measured at around 50% in surveys of usual medical care. On data obtained abroad: correlation with improved monitoring INR monitoring the ACC decreases by a factor 3-4 morbidity and mortality associated with the use of VKA and thus allows a significant reduction in hospitalizations caused by adverse drug effects and thus health care costs. In France several ACC, have emerged since 1998. Ile de France since 2004, the ACC Ile-de-France called CREATIF (Centre for Reference and Education antithrombotic Ile de France). Since its inception to date, has an active list of approximately 450 patients which monitors long-term anticoagulant treatment. The question of benefit of such a structure arises, is why this has been decided to establish a prospective randomized study to evaluate the benefit of the management of oral anticoagulant treatment by CREATIF with respect to usual medical care in terms of time in therapeutic INR range. This study of usual care, witch aims to assess two types of management of anticoagulant therapy, does not alter the type of anticoagulant therapy nor its duration. The overall medical care of patient and his care pathway will also remain unchanged. The study Randomized GP investigators, is open, prospective, is concerning primary medical care (independent central randomization). Primary care investigators are GPs managing patients treated by VKAs. They were recruited in a list of GPs working with CREATIF or through several physicians networks (North Paris Health Network, ARES 92, GP Department of Paris VII university, GP Department of Paris West). CREATIF, investigators will be usual physicians working at the anti-coagulation clinic. The aim of the study is to compare the management of patients treated with VKA by the CREATIF versus their management in primary care. Therefore, the evaluation criterion is the time in therapeutic INR range. During 6 months randomized in 2 arms: GPs versus CREATIF; During the next 6 months following the reversal mode of management is to determine the existence of prolonged benefit by one followed by CREATIF after returning to his usual medical care. The investigators will also collect the retrospective 6 months INR.A retrospective study, prospective, open and multicenter with direct individual benefit. Prospective study conducted in cross-over: anticoagulant therapy for each patient will be followed by six months CREATIF then by his GP or vice VERSA.Primary analysis: comparing the two types of monitoring parallel group after randomization: Group A in Phase 1 versus Group B in Phase 1. Primary endpoint: percentage of time in therapeutic INR range.

The main requirements of the commitment to the inclusion of GP will be:

To have a fax or email to communicate with the CREATIF To transmit its coordinated to CREATIF. Allow the TEC and the ARC to have access to medical records for establish the retrospectives records.

Support the CREATIF approach, by a letter signed sent to medical laboratories for INR values of the retrospective study.Patients treated by VKA: COUMADINE or PREVISCAN

ELIGIBILITY:
Inclusion Criteria:

INCLUSION CRITERIA OF DOCTORS:

General Physicians in the city and have agreed to participate in the study by signing an undertaking.

INCLUSION CRITERIA OF PATIENT:

* Patient has not expressed its opposition to the use of data as part of research
* Patient man or woman whose age is ≥ 18 years
* Patients whose condition requires treatment by VKAs PREVISCAN® or COUMADINE® with an INR target in areas following: 2 to 3 (target 2.5), 2.5 to 3.5 (target 3) or 3 to 4.5 (target 3.75)
* Patient for which the oral anticoagulant treatment had been prescribed and administered for at least 6 months
* Patient insured under Social Security

Exclusion criteria:

-Patient treated by SINTROM®

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2011-05; Primary Completion 2013-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Proportion of time in the therapeutic anticoagulation range ± 0.5 INR unit. | at 13 months
  INR goal according following areas:
  • 2 to 3 (target 2.5) / 2.5 to 3.5 (Target 3) / 3 to 4.5 (target 3.75). Anticoagulation quality was measured using percentage of time in therapeutic INR range (%TTR). Absolute difference of 10% of TTR, taking into account the published data showing a percentage of time in therapeutic INR range of about 50% with a standard deviation of around 23% in usual medical care.

SECONDARY OUTCOMES:
Reduce accidents and iatrogenic cost, which may be related to VKA (major haemorrhage and thrombosis). | at 13 months
Number of INR prescribed by the GP during usual medical care compared with the number of INR prescribed under Monitoring by the CREATIF | at 13 months
Score of education one month before and after the formation session | at 13 months

CONTACTS AND LOCATIONS:
Overall Officials: Ludovic DROUET, MD,PhD, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (2):
- France (2):
  - Service d'hématologie - Hôpital Lariboisière, Paris
  - 50, rue de la Justice, Paris